CLINICAL TRIAL: NCT06239337
Title: Evaluation of Xpert MTB/RIF Ultra in Stools and Urine to Improve Tuberculosis Diagnosis in Children
Status: Completed | Type: Observational
Sponsor: Medecins Sans Frontieres, Spain (Other)
Collaborators: Ministry of Health, Guinea-Bissau (Unknown); Ministry of Health, South Sudan (Unknown); Institute of Tropical Medicine, University of Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: MSF18115
Record Dates: First submitted 2024-01-15; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Tuberculosis; Pediatric Infectious Disease
Keywords: Pediatric TB; Xpert MTB/RIF Ultra; Stools; Urine
MeSH Terms: conditions — Tuberculosis | interventions — Defecation; Urination

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Biospecimen Retention: Samples With DNA — Respiratory, extrapulmonary, stools and urine specimens for Xpert MTB/RIF Ultra. Urine for TB LAM.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Xpert MTB/RIF Ultra in stools and urine — All children with presumptive TB had at least 1 sample collected of respiratory or extrapulmonary specimen (considered as gold standard) and 1 sample of stools and 1 sample of urine. All of them were analyzed with Xpert MTB/RIF Ultra.

SUMMARY:
Tuberculosis (TB) diagnosis in children is challenging in low and middle-income countries where access to TB culture and X-ray is limited. More than half cases of childhood TB remain undiagnosed every year. A delay in TB diagnosis can lead to an increase in preventable morbidity and mortality.

This study aims to provide evidence on the diagnostic accuracy of Xpert MTB/RIF Ultra in stools and urine for TB diagnosis in children.

DETAILED DESCRIPTION:
This multicentric cross-sectional study took place at Malakal hospitals from November 2019 to December 2023, and at Simão Mendes National Hospital between July 2019 and April 2020. Children with presumptive TB underwent clinical and laboratory evaluation.

Study Population, Clinical, and Laboratory procedures Children 6 months to 15 years were considered presumptive TB cases if they showed persistent cough for more than 2 weeks, unexplained fever for more than 1 week or signs of extrapulmonary TB such as: gibbous deformity of the spine, lymphadenopathy, subacute meningitis, distended abdomen with ascites, diarrhoea for more than two weeks, painless enlarged joints, or pleural effusion.

Presumptive TB cases were also identified after a week of inpatient admission, characterized by low weight gain despite nutritional treatment, persistent pneumonia or cough despite adequate antibiotic therapy, persistent fever (>38ºC), and persistent or aggravated fatigue. Patients were screened for TB based on their medical history and clinical presentation, including TB contacts, past TB treatment or known HIV infection; physical examination was conducted in all patients and included relevant anthropometrics (Mid-Upper-Arm Circumference (MUAC), Weight-for-height z scores (WHZ) and/or body mass index (BMI) for age z scores). All patients with unknown HIV status were tested for HIV and were tested for at least one pulmonary or extrapulmonary sample (considered as gold standard), and one stool and one urine samples.

All patients underwent a diagnostic evaluation and were included in three different categories: Confirmed TB (patients who had an Xpert MTB/RIF Ultra positive in one of the samples); Unconfirmed TB (clinical TB diagnosis without microbiological confirmation); Unlikely TB (alternative diagnosis with adequate response to alternative treatments, and TB treatment not started).

Respiratory samples included naso-pharyngeal aspirate, gastric lavage, or spontaneous sputum; extrapulmonary samples included lymph node puncture, pus aspirate, and ascetic, pleural, or cerebrospinal fluids. Stools and urine were collected from all patients as well. All specimens were kept between 2 and 8ºC until processed, which was done within 24 hours. Xpert MTB/RIF Ultra was performed in all collected sample.

In Malakal, MSF supported the TB program in collaboration with the Ministry of Health (MoH) all along the study. In Bissau, all results were communicated to MoH who were responsible for treatment initiation.

ELIGIBILITY:
Inclusion Criteria:

* Any child from 6 months of life to 15 years old
* TB suspected according to diagnostic criteria
* Informed consent provided by legal responsible or companion

Exclusion Criteria:

* Patients who have received TB treatment for > 1 day in the last 3 months
* Patients not producing stools or urine during period of admission and prior to starting TB drugs

Ages: 6 Months to 15 Years | Sex: All
Age Groups: Child
Study Population: The research population are children with presumptive TB at Malakal hospitals (South Sudan) at Simão Mendes National Hospital (Guinea-Bissau).
Sampling Method: Non-Probability Sample
Enrollment: 563 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
To determine the sensitivity and specificity of Xpert MTB/RIF Ultra in stool and urine samples in presumptive TB pediatric cases in comparison to Xpert MTB/RIF Ultra in respiratory/extrapulmonary sample | Through study completion, up to 60 months
  To determine the sensitivity and specificity of Xpert MTB/RIF Ultra in stool and urine samples in presumptive TB pediatric cases in comparison to Xpert MTB/RIF Ultra in respiratory/extrapulmonary sample

SECONDARY OUTCOMES:
To determine sensitivity and specificity of Xpert MTB/RIF Ultra in stool and urine samples in subpopulations: HIV/not HIV, SAM/no SAM, <5 years old vs. 5 or more years old. | Through study completion, up to 60 months
  To determine sensitivity and specificity of Xpert MTB/RIF Ultra in stool and urine samples in subpopulations: HIV/not HIV, SAM/no SAM, <5 years old vs. 5 or more years old.
To determine the added diagnostic yield of Xpert MTB/RIF Ultra in stool and urine samples when gold standard is negative | Through study completion, up to 60 months
  To determine the added diagnostic yield of Xpert MTB/RIF Ultra in stool and urine samples when gold standard is negative

CONTACTS AND LOCATIONS:
Overall Officials: Laura Moretó Planas, MD, Principal Investigator — MSF OCBA
Locations (2):
- Simao Mendes hospital, Bissau, Guinea-Bissau
- Malakal hospital, Malakal, Upper Nile, South Sudan

IPD SHARING:
Plan to Share IPD: No
This study will follow MSF data protection policy and IPD will be shared under request to Medical Director.

REFERENCES:
- [Background] Jenkins HE, Yuen CM, Rodriguez CA, Nathavitharana RR, McLaughlin MM, Donald P, Marais BJ, Becerra MC. Mortality in children diagnosed with tuberculosis: a systematic review and meta-analysis. Lancet Infect Dis. 2017 Mar;17(3):285-295. doi: 10.1016/S1473-3099(16)30474-1. Epub 2016 Dec 8. PMID 27964822
- [Background] POSEE Info Note_Pediatric TB diagnosis_Final_17.6.2021.pdf. Taskforce PTOaSEEP. Summary guidance for Microbiological and Clinical Diagnosis of pulmonary tuberculosis among Children: Pediatric TB Operational and Sustainability Expertise Exchange (POSEE) Taskforce, 2021.
- [Background] Dodd PJ, Prendergast AJ, Beecroft C, Kampmann B, Seddon JA. The impact of HIV and antiretroviral therapy on TB risk in children: a systematic review and meta-analysis. Thorax. 2017 Jun;72(6):559-575. doi: 10.1136/thoraxjnl-2016-209421. Epub 2017 Jan 23. PMID 28115682
- [Background] WHO consolidated guidelines on tuberculosis: Module 5: Management of tuberculosis in children and adolescents [Internet]. Geneva: World Health Organization; 2022. Available from http://www.ncbi.nlm.nih.gov/books/NBK579387/ PMID 35404556
- [Background] Kay AW, Ness T, Verkuijl SE, Viney K, Brands A, Masini T, Gonzalez Fernandez L, Eisenhut M, Detjen AK, Mandalakas AM, Steingart KR, Takwoingi Y. Xpert MTB/RIF Ultra assay for tuberculosis disease and rifampicin resistance in children. Cochrane Database Syst Rev. 2022 Sep 6;9(9):CD013359. doi: 10.1002/14651858.CD013359.pub3. PMID 36065889
- [Background] Atherton RR, Cresswell FV, Ellis J, Kitaka SB, Boulware DR. Xpert MTB/RIF Ultra for Tuberculosis Testing in Children: A Mini-Review and Commentary. Front Pediatr. 2019 Feb 28;7:34. doi: 10.3389/fped.2019.00034. eCollection 2019. PMID 30873392
- [Background] Vessiere A, Font H, Gabillard D, Adonis-Koffi L, Borand L, Chabala C, Khosa C, Mavale S, Moh R, Mulenga V, Mwanga-Amumpere J, Taguebue JV, Eang MT, Delacourt C, Seddon JA, Lounnas M, Godreuil S, Wobudeya E, Bonnet M, Marcy O. Impact of systematic early tuberculosis detection using Xpert MTB/RIF Ultra in children with severe pneumonia in high tuberculosis burden countries (TB-Speed pneumonia): a stepped wedge cluster randomized trial. BMC Pediatr. 2021 Mar 20;21(1):136. doi: 10.1186/s12887-021-02576-5. PMID 33743621
- [Background] Kabir S, Rahman SMM, Ahmed S, Islam MS, Banu RS, Shewade HD, Thekkur P, Anwar S, Banu NA, Nasrin R, Uddin MKM, Choudhury S, Ahmed S, Paul KK, Khatun R, Chisti MJ, Banu S. Xpert Ultra Assay on Stool to Diagnose Pulmonary Tuberculosis in Children. Clin Infect Dis. 2021 Jul 15;73(2):226-234. doi: 10.1093/cid/ciaa583. PMID 32421765
- [Background] Sun L, Liu Y, Fang M, Chen Y, Zhu Y, Xia C, Jia J, Quan S, Wang Y, Tian X, Shi Y, Duan L, Shi X, Liao Q, Wan C, Shen A. Use of Xpert MTB/RIF Ultra assay on stool and gastric aspirate samples to diagnose pulmonary tuberculosis in children in a high-tuberculosis-burden but resource-limited area of China. Int J Infect Dis. 2022 Jan;114:236-243. doi: 10.1016/j.ijid.2021.11.012. Epub 2021 Nov 10. PMID 34774781
- [Derived] Moreto-Planas L, Mahajan R, Fidelle Nyikayo L, Ajack YBP, Tut Chol B, Osman E, Sangma M, Tobi A, Gallo J, Biague E, Goncalves R, Rocaspana M, Medina C, Camara M, Flevaud L, Ruby LC, Belard S, Sagrado MJ, Molina I, Llosa AE. Xpert-Ultra Assay in Stool and Urine Samples to Improve Tuberculosis Diagnosis in Children: The Medecins Sans Frontieres Experience in Guinea-Bissau and South Sudan. Open Forum Infect Dis. 2024 May 2;11(5):ofae221. doi: 10.1093/ofid/ofae221. eCollection 2024 May. PMID 38798893

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT06239337/Prot_SAP_ICF_000.pdf